CLINICAL TRIAL: NCT04722627
Title: A First-in Human, Randomized, Double-blind, Placebo Controlled Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AT-752 in Healthy Subjects
Brief Title: Study of AT-752 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-02A-001
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — AT-752

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- AT-752 250 mg single dose (Experimental): AT-752 administered orally, 250 mg on Day 1
  Interventions: Drug: AT-752
- Placebo -single dose (Placebo Comparator): Matching placebo administered orally on Day 1
  Interventions: Drug: Placebo
- AT-752 500 mg single dose (Experimental): AT-752 administered orally, 500 mg single doses on Day 1 and Day 7
  Interventions: Drug: AT-752
- Placebo- single dose (Placebo Comparator): Matching placebo administered orally on Day 1 and Day 7
  Interventions: Drug: Placebo
- AT-752 1000 mg single dose (Experimental): AT-752 administered orally, 1000 mg single dose on Day 1
  Interventions: Drug: AT-752
- Placebo - single dose (Placebo Comparator): Matching placebo administered orally on Day 1
  Interventions: Drug: Placebo
- AT-752 1500 mg single dose (Experimental): AT-752 administered orally, 1500 mg single dose on Day 1
  Interventions: Drug: AT-752
- Placebo: single dose (Placebo Comparator): Matching placebo administered orally on Day 1
  Interventions: Drug: Placebo
- AT-752 - 1000 mg QD multiple doses (Experimental): AT-752 - administered orally, 1000 mg once daily (QD) for 7 days
  Interventions: Drug: AT-752
- Placebo - Administered once daily (QD) (Placebo Comparator): Matching placebo administered orally once daily (QD) for 7 days
  Interventions: Drug: Placebo
- AT-752 - 750 mg twice daily (BID) (Experimental): AT-752 administered orally, 750 mg twice daily (BID) for 4 days plus one dose on Day 5.
  Interventions: Drug: AT-752
- Placebo - Administered twice daily (BID) (Placebo Comparator): Matching placebo administered orally twice daily (BID) for 4 days plus one dose on Day 5.
  Interventions: Drug: Placebo
- AT-752 - 750 mg three times daily (TID) (Experimental): AT-752 administered orally, 750 mg three times daily (TID) for 4 days plus one dose on Day 5.
  Interventions: Drug: AT-752
- Placebo - Administered TID (Placebo Comparator): Matching placebo administered orally (TID) for 4 days plus one dose on Day 5.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AT-752 — Parallel Assignment
  Arms: AT-752 - 1000 mg QD multiple doses; AT-752 - 750 mg three times daily (TID); AT-752 - 750 mg twice daily (BID); AT-752 1000 mg single dose; AT-752 1500 mg single dose; AT-752 250 mg single dose; AT-752 500 mg single dose
Drug: Placebo — Parallel Assignment
  Arms: Placebo - Administered TID; Placebo - Administered once daily (QD); Placebo - Administered twice daily (BID); Placebo - single dose; Placebo -single dose; Placebo- single dose; Placebo: single dose

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) of AT-752 in healthy subjects

DETAILED DESCRIPTION:
A First-in Human, Randomized, Double-blind, Placebo controlled Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AT-752 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) of 18-29 kg/m2
2. Must agree to use protocol-specified methods of contraception
3. Negative pregnancy test
4. Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Abuse of alcohol or drugs
3. Use of other investigational drugs within 30 days of dosing
4. Other clinically significant medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Proportions (active vs. Placebo) of subjects experiencing treatment-emergent adverse events | Day 6 for single dose or Day 12 for multiple dose
Pharmacokinetics (PK) of AT-752 of single and multiple ascending oral doses | Day 1 for subjects receiving a single fasted dose; Days 1 and 7 for subjects receiving multiple doses
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of AT-752 of single and multiple ascending oral doses | Day 1 for subjects receiving a single fasted dose; Days 1 and 7 for subjects receiving multiple doses ]
  Area under the concentration-time curve (AUC)
Effect of food on Pharmacokinetics (PK) of AT-752 of a single oral dose | Day 1 for subjects receiving a single fed dose]
  Maximum plasma concentration (Cmax)
Effect of food on Pharmacokinetics (PK) of AT-752 of a single oral dose | Day 1 for subjects receiving a single fed dose ]
  Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou X-J, Lickliter J, Montrond M, Ishak L, Pietropaolo K, James D, Belanger B, Horga A, Hammond J. First-in-human trial evaluating safety and pharmacokinetics of AT-752, a novel nucleotide prodrug with pan-serotype activity against dengue virus. Antimicrob Agents Chemother. 2024 May 2;68(5):e0161523. doi: 10.1128/aac.01615-23. Epub 2024 Mar 25. PMID 38526047